CLINICAL TRIAL: NCT06289738
Title: Problem Analysis Based on the International Classification of Functioning, Disability and Health in Patients With Takayasu Arteritis
Brief Title: ICF in Takayasu Arteritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, Assistant Professor, Uşak University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICF in Takayasu Arteritis
Record Dates: First submitted 2024-02-24; First posted 2024-03-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Takayasu Arteritis patients between the ages of 18-65
  Interventions: Other: ICF

INTERVENTIONS:
Other: ICF — Matching the answers given to the question set consisting of 6 open-ended questions with ICF

SUMMARY:
The aim was to analyze the problem in patients with Takayasu Arteritis based on the International Classification of Functioning, Disability and Health.The sample of our study will consist of individuals between the ages of 18-65 who have been diagnosed with Takayasu Arteritis by rheumatologists and are followed by Pamukkale University Rheumatology Clinic.

ELIGIBILITY:
Inclusion Criteria:-Being between the ages of 18-65

* Volunteering to participate in the study
* Being diagnosed with Takayasu Arteritis by a rheumatologist

Exclusion Criteria:- Having another disease that affects your physical condition

* Having cognitive impairment that makes it difficult to cooperate
* Being pregnant
* Having a neurological disease
* Having had any surgery in the last year
* Having another concurrent rheumatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
6 open-ended questions | 25 minutes
  ICF

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Gur Kabul, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No